CLINICAL TRIAL: NCT07003971
Title: Investigation of the Effectiveness of Social Media-Based Support in Developing Healthy Lifestyle Behaviors in Pregnancy
Brief Title: The Effect of Social Media Support on Healthy Lifestyle Behaviours
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ozlem TAS, PhD Candidate, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/177
Record Dates: First submitted 2025-05-03; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Social Media in Developing Healthy Lifestyle Behaviours in Pregnant Women
Keywords: pregnant women, pregnancy, social media, healthy lifestyle
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The research will be conducted in a prospective pre-test, post-test randomised controlled experimental research design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- social media participants (Experimental): In addition to routine care and counseling, pregnant women in the experimental group will be offered support to develop healthy lifestyle behaviors through Instagram.
  * Creating and naming the Instagram account for the presentation of the programme planned to create Healthy Lifestyle Behaviours,
  * Creating programme contents for developing Healthy Lifestyle Behaviours,
  * Transferring the content prepared to develop Healthy Lifestyle Behaviours to the Instagram platform,
  * Sharing the training on developing Healthy Lifestyle Behaviours with pregnant women in the experimental group via Instagram and trying to create these behaviours in pregnant women,
  * It is planned to reveal the effect of the content aimed at developing Healthy Lifestyle Behaviours on the acquisition of healthy living habits of pregnant women by presenting them through Instagram with a randomised controlled study.
  Interventions: Behavioral: counselling
- Control (Other): The control group will not be trained in Instagram, but will be provided with standardised medical care established by the Turkish Ministry of Health during the follow-up period.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: counselling — After the participants in the experimental group signed the 'Informed Consent Form', the Instagram addresses actively used by the pregnant women participating in the study will be taken, the Instagram account created by the researcher will be shared with the pregnant women in the experimental group, the participants will be ensured to follow the Instagram address created by the researcher and join the Instagram DM group. After the participation to the platform is completed, the visibility of the participants in the account will be checked. After the visibility of all participants is ensured, pre-tests created in Google Forms and uploaded to WhatsApp and Instagram DM group will be applied.
  Arms: social media participants
Other: Control — After the 'Informed Consent Form' is signed by the pregnant women in the control group, the telephone numbers of the participants will be taken and recorded in the directory. Participants will also be asked to save the researcher's phone number. After being registered in the phone book, questionnaires and scales will be shared via WhatsApp and asked to answer the pre-tests prepared in Google Forms. Pregnant women who answer will be asked to return with a WhatsApp message in the form of 'I answered' or 'I sent'. The control group will not be trained on Instagram, but will be provided with standardised medical care established by the Turkish Ministry of Health during the follow-up period.
  Arms: Control

SUMMARY:
The aim of this study is to examine the effectiveness of a programme to improve healthy lifestyle behaviours based on the Health Belief Model to be offered through Instagram, a social media platform. For this purpose, it is aimed to produce content containing accurate and evidence-based information for pregnant women on social media, to ensure that pregnant women can access the right information quickly and easily, to adopt healthy lifestyle behaviours, to test the effectiveness of the social media platform for the adoption of healthy lifestyle behaviours and to contribute to the formation of a healthier family and society in the long term. In addition, this study is aimed to create a model for the midwifery profession to benefit from the new opportunities created by internet technology outside the clinical field in service delivery.

The population of the study will consist of women with primiparous pregnancies in the first and second trimester. Women who agree to participate in the study will be randomly assigned to the experimental and control groups. In addition to routine care and counselling, pregnant women in the experimental group will receive support for developing healthy lifestyle behaviours through Instagram, while the control group will receive only standard pregnancy care and counselling services approved by the Ministry of Health.

General Hypothesis of the Study:

H1: The Healthy Lifestyle Behaviours development programme offered through the social media platform Instagram is effective in providing a positive development on healthy lifestyle behaviours in pregnant women.

DETAILED DESCRIPTION:
Maternal health covers women's health during pregnancy, childbirth and the postnatal period. Despite significant progress over the last two decades, 287,000 women are reported to die during pregnancy, childbirth and the postnatal period in 2020. Adopting healthy lifestyle habits from pre-pregnancy to the postnatal period is crucial for healthy pregnancies and the prevention of diseases that can occur during pregnancy. Pregnant women are advised to adopt healthy eating habits, consume adequate nutrients, balance the body's extra demands and maintain physical activity to maintain good health and prevent excessive weight gain. The World Health Organisation warns pregnant women about nutrition, physical activity, stress management and avoiding toxic substances. High-quality evidence shows that diet, exercise or both interventions can significantly reduce the risk of excessive pregnancy weight gain compared with routine care. These interventions may reduce maternal hypertension, neonatal respiratory distress syndrome, caesarean section, macrosomia. Today, a large part of our lives is dominated by mobile phones, computers and household appliances that operate over the Internet. In this way, people can communicate with each other and transfer information to each other without time and space barriers. Social media, defined as online networking sites that enable Internet users to communicate through activities such as content sharing and personal comments, has become a widely used term for sharing information and ideas on the Internet or mobile platforms. The literature shows that the use of social media has become widespread in pregnancy care. In a meta-analysis of fifteen randomised controlled trials, social media and mobile health applications were found to be effective in supporting maternal physical health in pregnant women in conditions such as weight management, gestational diabetes control, asthma control. At the same time, it has been observed that it improves maternal mental health and increases women's level of knowledge about the pregnancy process.

With the current study, it is aimed to implement the Healthy Lifestyle Behaviour Development Programme to be created based on the Health Belief Model in pregnant women through the social media platform, which is frequently used today, and to contribute to the development of mother-baby health by providing pregnant women with instant and easy access to the right information.

ELIGIBILITY:
Inclusion Criteria:

* First and second trimester pregnancy
* 18-49 years old
* With a singleton pregnancy
* Able to use web and mobile devices
* Has an account of the determined social media platform and actively uses it
* Can read and write Turkish
* Pregnant women with regular internet access were included in the inclusion criteria of this study.

Exclusion Criteria:

* Has a psychiatric problem that prevents communication
* Have a serious pre-pregnancy condition (heart disease, kidney disease or other chronic disease)
* Previously used a similar programme or app to change healthy lifestyle habits
* Risky pregnancies (heart disease, kidney disease or other chronic diseases)

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The group to be trained during their pregnancy consists of women.
Enrollment: 96 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Developing healthy lifestyle behaviours in pregnant women | 8 weeks
  To ensure the formation of healthy lifestyle behaviours in pregnant women It was developed by Walker et al. (1996) and adapted into Turkish by Bahar et al. (2008). Scale; Health Responsibility (3,9,15,21,27,33,39,45,51), Physical Activity (4,10,16,22,28,34,40,46), Nutrition (2,8,14,20,26,32,38,44,50), Spiritual Development (6,12,18,24,30,36,42,48, 52), Interpersonal Relationships (1,7,13,19,25,25,31,37,43,49), Stress Management (5,11,17,23,29,35,41,47). The scale was used to measure healthy lifestyle behaviors and validity and reliability studies were conducted. The Cronbach Alpha coefficient of the scale is .92 and has a high degree of reliability. The reliability coefficients of the sub-dimensions of the scale were found to be; Health responsibility .77, Physical Activity .79, Nutrition .68, Spiritual Development .79, Interpersonal Relations .80, Stress Management .64. Increasing scores in the total scale and sub-dimensions indicate a positive attitude towards healthy lifestyle beh
Pregnant women who participate in a program to improve healthy lifestyle behaviors offered through Instagram will have better sleep quality. | 8 weeks
  Since there is no section evaluating sleep in the Healthy Lifestyle Behaviors Scale, it was found appropriate to use a separate scale. The DSM-5 Sleep Disorder Scale was developed to measure the severity of sleep problems according to DSM-5 criteria (Yu et al. 2012; Yüzeren et al. 2017; https://www.psychiatry.org). The scale, also known as PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disorder Scale Short Form, is a well-structured measurement tool (Yüzeren et al. 2017; Ravyts et al. 2021) and has been used in pregnant women (Haas et al. 2016; Bei et al. 2019). The validity and reliability study of the DSM-5 Sleep Disorder Scale Turkish Form (PROMIS-Sleep Disorder Scale-Short Form) (ANNEX-6), which is planned to be used in this study, was conducted by Yüzeren et al. in 2017. The scale, which is suitable for adults, is filled out by taking into account the sleep patterns and quality of people between the ages of 18-75 in the last seven days.
Pregnant women who participate in a program to improve healthy lifestyle behaviors offered through the Instagram platform may have a more positive attitude towards endocrine disruptors. | 8 weeks
  Endocrine Disruptors Attitude Scale (EDAS):
  Since the Healthy Lifestyle Behaviors Scale does not have a section evaluating the attitude towards endocrine disruptors, it was found appropriate to use a separate scale. The scale was developed by Miral et al (2022) to determine adults' attitudes towards endocrine disruptors and consists of 21 items. The endocrine disruptors attitude scale has two sub-dimensions: consumer behavior and nutrition and hygiene. The consumer behavior sub-dimension consists of 11 items in total, including items numbered 1,2,7,8,9,9,10,10,11,12,12,13,18,21. The nutrition and hygiene sub-dimension consists of 10 items in total, including items numbered 3,4,5,6,14,15,16,17,19,20. The scale was prepared as a five-point Likert-type scale as "Strongly agree", "Agree", "Neutral", "Disagree", "Strongly disagree". There are no reverse items in the scale. The highest score to be obtained from the scale, which has no cut-off value, is 105 and the lowest score is 21.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Özcan, Prof. Dr., Study Director — Istanbul Univercity-Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stephenson J, Heslehurst N, Hall J, Schoenaker DAJM, Hutchinson J, Cade JE, Poston L, Barrett G, Crozier SR, Barker M, Kumaran K, Yajnik CS, Baird J, Mishra GD. Before the beginning: nutrition and lifestyle in the preconception period and its importance for future health. Lancet. 2018 May 5;391(10132):1830-1841. doi: 10.1016/S0140-6736(18)30311-8. Epub 2018 Apr 16. PMID 29673873
- [Background] Oli N, Vaidya A, Pahkala K, Eiben G, Krettek A. Knowledge, attitude and practice on diet and physical activity among mothers with young children in the Jhaukhel-Duwakot Health Demographic Surveillance Site, Nepal. PLoS One. 2018 Jul 9;13(7):e0200329. doi: 10.1371/journal.pone.0200329. eCollection 2018. PMID 29985946
- [Background] Katenga-Kaunda LZ, Kamudoni PR, Holmboe-Ottesen G, Fjeld HE, Mdala I, Shi Z, Iversen PO. Enhancing nutrition knowledge and dietary diversity among rural pregnant women in Malawi: a randomized controlled trial. BMC Pregnancy Childbirth. 2021 Sep 22;21(1):644. doi: 10.1186/s12884-021-04117-5. PMID 34551744
- [Background] Hojeij B, Schoenmakers S, Willemsen S, van Rossem L, Dinnyes A, Rousian M, Steegers-Theunissen RP. The Effect of an eHealth Coaching Program (Smarter Pregnancy) on Attitudes and Practices Toward Periconception Lifestyle Behaviors in Women Attempting Pregnancy: Prospective Study. J Med Internet Res. 2023 Jan 31;25:e39321. doi: 10.2196/39321. PMID 36719733
- See also: World Health Organization (WHO), 2022a. Be Healthy Mobile. — https://www.who.int/initiatives/behealthy/.